CLINICAL TRIAL: NCT06295965
Title: Clonal Hematopoiesis and Therapy-Emergent Myeloid Neoplasms in Patients With Cancers (CHANCES)
Brief Title: Clonal Hematopoiesis and Therapy-Emergent Myeloid Neoplasms in Patients With Cancers, CHANCES Study
Status: Recruiting | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: RG1123813; NCI-2023-10315 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0020162 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA272594 (NIH)
Record Dates: First submitted 2024-02-06; First posted 2024-03-06 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Recurrent Malignant Solid Neoplasm; Clonal Cytopenia of Undetermined Significance; Clonal Hematopoiesis; Idiopathic Cytopenia of Undetermined Significance; Non-Neoplastic Hematopoietic and Lymphoid Cell Disorder; Ovarian Carcinoma; Myeloid Neoplasm Post Cytotoxic Therapy
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients undergo blood sample collection and complete surveys on study. Patients' medical records are also reviewed.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study is being done to investigate clonal hematopoiesis and therapy-emergent myeloid neoplasms in patients with ovarian or other solid cancers. Researchers want to identify risk factors for developing these blood cancers as well as if there is/are a genetic/environmental component(s) to developing blood cancer.

DETAILED DESCRIPTION:
OUTLINE: This is an observational study.

Patients undergo blood sample collection and complete surveys on study. Patients' medical records are also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have or have had ovarian, peritoneal, or fallopian tube carcinoma who have a life expectancy of greater than 6 months and:

  * Have completed or plan to complete at least 5 cycles of platinum-based chemotherapy

OR

* Subjects who have or have had a solid tumor diagnosis and any of the following:

  * At least 4 months of exposure to a PARP inhibitor
  * Diagnosis of a blood disorder including, but not limited to, clonal hematopoiesis of indeterminate potential, cytopenia of unknown significance, or therapy-related myeloid neoplasm

Exclusion Criteria:

* Individuals with a life expectancy of less than 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who have had ovarian, peritoneal, or fallopian tube cancer and have completed or plan to complete at least 5 cycles of platinum-based chemotherapy or subjects who have had a solid tumor diagnosis and have received at least 4 months of PARP inhibitor and/or been diagnosed with a blood disorder.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine the correlation between baseline TP53m VAF in blood with CH expansion in OC patients | Through study completion, up to 5 years
Identify risk of TMN for OC survivors with and without TP53m CH treated with platinum chemotherapy and PARP inhibitors | Through study completion, up to 5 years
  Measurement Tool: will measure by BM biopsy confirmation done by local hematologist
Define the trajectories of clonal evolution and mechanisms of transformation from non-cancerous TP53m to TMN | Through study completion, up to 5 years
  Measurement Tool: the variant allele fraction of the blood clone

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Swisher, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No